CLINICAL TRIAL: NCT04346966
Title: The Effectiveness of Video-Based Exercises in Young Adults Under Social Isolation Process Due to Coronavirus
Brief Title: The Effectiveness of Video-Based Exercises in Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, Yasemin Çırak, Physiotherapist, PhD, Associate Professor, Istinye University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 001
Record Dates: First submitted 2020-04-13; First posted 2020-04-15 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Social Isolation; Exercise; Healthy
Keywords: Physical Activity; COVID-19; Young adults
MeSH Terms: conditions — Social Isolation; Motor Activity; COVID-19

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): The group to which the exercise videos consisting of aerobic and strengthening exercises will be applied.
  Interventions: Other: Study Group
- Control Group (No Intervention): The control group where only the evaluations will be made and information about the benefits of exercise will be given.

INTERVENTIONS:
Other: Study Group — Video Based Exercises 64 young adults aged 18-40, who are socially isolated due to coronavirus, will be included in this group. A video-based exercise protocol was created for individuals to participate in the study. Each exercise session is planned as 30 minutes 7 days a week for 6 weeks. The protocol was planned to start with warm-up exercises and end with cooling exercises. The exercise protocol has also been determined as a combination of aerobic exercises, strengthening and posture exercises. Individuals will be classified at 4 levels according to their physical activity levels and will be shared with volunteers according to their level of exercise. Volunteers will be evaluated before and after 6 weeks of exercise.
  Arms: Study Group

SUMMARY:
In December 2019, the new coronavirus pneumonia (COVID-19) exploded in Wuhan (Hubei, China) and spread rapidly from one city to the whole world. This virus resulted in a total of 1679720 confirmed cases and 101734 deaths worldwide. All countries in the world are taking some precautions to prevent the spread of this epidemic disease, which World Health Organization (WHO) declared as "epidemic". Staying home and social isolation are among these precautions. For this purpose, it began to implement the curfew for all individuals on 10 March 2020, Turkey. However, not leaving the house and social isolation bring about the limitation of physical activity. Physical activity (PA) is defined as anybody's movement produced by WHO by contraction of skeletal muscles. Studies investigating the relationship between social isolation and health behavior report consistent findings. Individuals with smaller social networks report less healthy diets, excessive alcohol consumption, and less physical activity. Traditional exercises; It takes place outdoors in gyms or rehabilitation centers. However, with the increase in the time we spent at home due to the coronavirus (COVID-19) epidemic, technologies have been used as an alternative method. Home-based exercise programs are also a viable solution to prevent various health problems that may be encountered in this direction. The decrease in physical performance is associated with loss of muscle strength, low quality of life, emotionalization, comorbidity, premature death, and increased health costs. When today's conditions are evaluated, technology-supported education programs are effective in increasing motivation for physical support. The purpose of this study; To prevent the spread of the COVID-19 outbreak, to evaluate the physical activity levels of individuals between the ages of 18-40 who have social isolation due to the measures taken in our country and to investigate the effectiveness of their video-based exercises.

DETAILED DESCRIPTION:
Sedentary life invites various diseases. Especially cardiovascular diseases are the leading ones. Researches show that the rapid development of technology has pushed people to laziness and therefore to immobility. A sedentary lifestyle causes many serious health problems. Many diseases such as obesity and cardiovascular diseases, which are characterized as contemporary diseases, such as muscular weakness, postural disorder, and diabetes are more common in immobile and sedentary individuals.

We know that still life has some drawbacks. These may cause tissue injuries between the vertebrae and kyphosis, lordosis, scoliosis problems, respectively. It may also cause calcification in the lumbar vertebrae, disc problems, risk of sciatica, and an increase in excess adipose tissue under the skin. Again high blood cholesterol and triglyceride findings and blood sugar abnormalities may occur in the blood table. Of course, the susceptibility to high blood pressure, the loss of elasticity of the rib cage, low respiratory capacity, and the risk of coronary vascular disease may be uncertain. Still life can create weak abdomen and back muscles, posture disorder, digestive and excretion difficulties, postpartum drooping abdomen, hip slope abnormality, loss of strength, flexibility and functionality in all muscle and muscle groups, weight problem and formlessness. Also in skeleton structure; osteoporosis, calcification, joint problems, easy injury, weak body, easy sickness and recovery can be observed. All these diseases are serious health problems that can be encountered in individuals who do not exercise regularly. In many developed countries of the world, people have included sports in many compulsory habits such as eating, drinking, lying, education, and worship. This compulsory exercise is a lifelong activity in humans. People who make it compulsory to exercise will feel discomfort as soon as they do not.

At the moment, we know that the most valid method to protect against coronavirus is to stay at home. Many scientists are told that this virus protection is to strengthen the immune system through exercise, and that the weight problem can be eliminated with exercise due to staying at home all day long. Because, it is explained one by one that exercise will increase the body resistance of the people, children and adults will stay away due to movement from obesity, the skeletal-muscular system will be regular, and the social environment will make people healthier.

In addition, constant home, restricted mobility and freedom, limited sociability, decreased communication, increased social-physical distance with our loved ones, and decreased physical contact can make us more depressed, angry and anxious.

For all these reasons, the home quarantine process created due to the Corona virus necessitates exercise. We believe that this process can be managed in the most effective way with video exercise and information booklets in order to reduce inactivity in this process, which is left at home with the philosophy of life is movement, movement is life.

Science and technology have been developing since the day human beings existed. Technology; It is used in many fields such as education, health, communication, defense, industry and transportation. Technology has brought many benefits and a new perspective to the health sector as well as other fields. In this study, it was aimed to investigate the effects of the exercise program that we applied remotely with video-based exercises during the quarantine days on the parameters such as physical activity level, balance, endurance, sleep quality, depression, anxiety and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-40
* Being a healthy individual
* To have the ability to understand and apply written and verbal instructions in education videos and booklets.
* Being in the process of social isolation

Exclusion Criteria:

* Exercising regularly for the last 6 weeks
* Taking a break from sports due to sports injury
* Having a coronary risk factor or any chronic condition that we cannot deal with
* Having a neurological problem
* Clinical conditions such as infection, kidney failure, thyrotoxicosis that may affect exercise performance or aggregate with exercise

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 128 (Actual)
Dates: Start 2020-08-20 (Actual); Primary Completion 2020-10-20 (Actual); Study Completion 2020-11-20 (Actual)

PRIMARY OUTCOMES:
International Physical Activity Questionnaire (Short Form) | 2 weeks
  This questionnaire was developed to determine the physical activity levels of participants aged 15-65.
  International Physical Activity Questionnaire (IPAQ) allows to calculate the metabolic equivalent threshold (MET) by measuring the frequency, process and physical activity intensity level over the last seven days across all contexts and provides the amount of weekly physical activity. It is calculated as a weekly working hour (MET-hour / week). It divides people into physical activity groups based on frequency and intensity of physical activity. MET calculated accordingly can be classified as low, medium and high level.
Short Form-36 (SF-36) | 2 weeks
  Short Form-36 is a set of generic, coherent, and easily administered quality-of-life measures. These measures rely upon patient self-reporting and are now widely utilized by managed care organizations and by Medicare for routine monitoring and assessment of care outcomes in adult patients.It contains 36 items
The Pittsburgh Sleep Quality Index | 2 weeks
  The Pittsburgh Sleep Quality Index (PSQI) is an effective instrument used to measure the quality and patterns of sleep in the older adult. It differentiates "poor" from "good" sleep by measuring seven domains: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction over the last month. The client self rates each of these seven areas of sleep. Scoring of the answers is based on a 0 to 3 scale, whereby 3 reflects the negative extreme on the Likert Scale.
  A global sum of "5"or greater indicates a "poor" sleeper.
Distress Tolerance Scale | 2 weeks
  The Distress Tolerance Scale (previously Distress Tolerance Questionnaire, DTQ) is a 15 item self-report measure of emotional distress tolerance. Individuals select on a 1-5 likert scale
  (Strongly Disagree, Mildly Disagree, Feel Neutral, Mildly Agree, Strongly Agree) about each of the 16 statements about distress. There is one total scale, and only item 6 is reverse coded.
Beck Anxiety Inventory | 2 weeks
  The Beck Anxiety Inventory (BAI) is a 21-question multiple-choice self-report inventory that is used for measuring the severity of anxiety in children and adults. The questions used in this measure ask about common symptoms of anxiety that the subject has had during the past week (including the day you take it) (such as numbness and tingling, sweating not due to heat, and fear of the worst happening). It is designed for individuals who are of 17 years of age or older and takes 5 to 10 minutes to complete. The BAI contains 21 questions, each answer being scored on a scale value of 0 (not at all) to 3 (severely). Higher total scores indicate more severe anxiety symptoms.
Nottingham Health Profile | 2 weeks
  Nottingham Health Profile was created in England in 1985 to evaluate the quality of life-related to health. The Nottingham Health Profile is a general quality of life questionnaire that assesses the level of individuals health problems and how they affect their daily life activities.
Sit And Reach Test | 2 weeks
  The sit and reach test is a common measure of flexibility, and specifically measures the flexibility of the lower back and hamstring muscles. This test involves sitting on the floor with legs stretched out straight ahead. Shoes should be removed. The soles of the feet are placed flat against the box. Both knees should be locked and pressed flat to the floor - the tester may assist by holding them down. With the palms facing downwards, and the hands on top of each other or side by side, the subject reaches forward along the measuring line as far as possible. Ensure that the hands remain at the same level, not one reaching further forward than the other. After some practice reaches, the subject reaches out and holds that position for at one-two seconds while the distance is recorded. Make sure there are no jerky movements.
Shoulder Flexibility Test | 2 weeks
  The shoulder flexibility test is a simple evaluation of the flexibility and mobility of your shoulder joint. Also known as the reach test or the Apley back scratch test, it is used to assess the range of motion (ROM) of your shoulder, including flexion and extension.
Curl-Up Test | 2 weeks
  The objective of the Curl-Up Test is to assess the endurance of the athlete's abdominal muscles. This test requires to complete as many curl-ups as possible at a rate of minute.
Repetitive Squat Test | 2 weeks
  The objective of this test is to assesment of the leg strength. This test requires the participant to complete as many squats as possible with no rest.
Side Plank Test | 2 weeks
  The side plank test is typically a measure of core endurance and dictates that the subject brace themselves in a neutral and extended side lying position on the forearm with the shoulder directly above the elbow, whilst the top leg and trunk is raised and held for as long as possible.
Timed Up and Go Test | 2 weeks
  The Timed Up and Go test (TUG) is a simple test used to assess a person's mobility and requires both static and dynamic balance.[1]
  It uses the time that a person takes to rise from a chair, walk three meters, turn around, walk back to the chair, and sit down. Test completion time recorded.
Single Leg Stance Test | 2 weeks
  Single Leg Stance Test is used to measure static balance. The person is asked to stand on one leg for 60 seconds. The time it remains in balance is recorded. Contact of the leg in the air with any surface is considered unsuccessful. It is applied in two different ways: eyes open and eyes closed.

CONTACTS AND LOCATIONS:
Locations (1):
- İstinye University, Istanbul, Turkey (Türkiye)